CLINICAL TRIAL: NCT06168838
Title: Anticoagulant-associated Intracranial Hemorrhage: Patient Characteristics and Outcomes From National Institute of Neurology and Neurosurgery Manuel Velasco: Single-Center Observational Study
Brief Title: Anticoagulant-associated Intracranial Hemorrhage
Acronym: AAIHINNN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Vanessa Cano, Principal Investigator, El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Other Study IDs: INNN-DI-CI-271-2023
Record Dates: First submitted 2023-09-01; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Anticoagulant-induced Bleeding; Intracranial Hemorrhages
Keywords: Anticoagulants; Intracranial hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anticoagulant — Know the casuistry of spontaneous intracranial hemorrhages and secondary to the use of both oral and parenteral anticoagulants
  Other Names: intracranial hemorrhage

SUMMARY:
Oral anticoagulant therapy, including factors Xa and 2a inhibitors has become more popular in recent years due to its efficacy and convenience in preventing thrombotic events and reducing the risk for stroke in patients with rosk factors (e.g. atrial fibrillation, deep venous thrombosis, pulmonary embolism). These drugs have replaced traditional therapies such as warfarin, which requires frequent dose adjustments and control blood samples. Warfarin also has a higher risk of bleeding events.

Many patients with atrial fibrillation, particularly old patients and those with comorbidities may have trouble achieving the dose and control requirements for warfarin therapy. On the other hand, Direct Oral Anticoagulant therapies do not require a close monitorization and have a lower risk of bleeding events, which makes them a more attractive option for many patients.

There is solid evidence behind the efficacy and safety of Direct Oral Anticoagulant therapies. Multiple clinical trials have demonstrated that Factor Xa inhibitors like rivaroxaban and apixaban are as effective as warfarin in preventing blood clots and reducing stroke risk in patients living with atrial fibrillation.

These challenges remark the need for new research that can improve our comprehension about the risk of bleeding associated to anticoagulant therapies and develop novel and more effective strategies for minimizing this risk.

Hence, an observational analysis about anticoagulant-associated intracranial hemorrhage may help identifying its incidence and prevalence, as well as treatment patterns and identifying any patient with risk factors linked to these events.

This information can be used to improve patient outcomes and guide future research.

Work Hypothesis: The majority of intracranial hemorrhage events are associated with heparin, low molecular weight heparin and warfarin instead of Factor Xa inhibitors or direct thrombin inhibitors. Nevertheless, the growing use in recent years of factor Xa inhibitors can increase the number of this therapy related bleeding events.

DETAILED DESCRIPTION:
Study observational. The total number of subjects for this study will be determined by the number of patients with intracranial bleeding associated with anticoagulant therapy on the clinical records.

Primary objective: To identify the incidence and prevalence of intracranial bleeding events associated to oral anticoagulant therapy including vitamin k antagonists, factor Xa inhibitors and factor 2a inhibitors.

Secondary objective:

* To identify mortality related to intracranial bleeding associated with oral anticoagulant therapy, including vitamin K antagonists, factor Xa inhibitors and factor 2a inhibitors.
* To identify patients´ characteristics correlated with intracranial hemorrhage associated with oral anticoagulants.
* To identify treatment patterns: anticoagulant-associated intracranial bleeding management, including clinical, pharmacological, surgical, and interventional treatments, as well as procoagulant therapies.

Sample size Justification / Statistical Analysis: Non probabilistic, incidental reasoned selection.

The sample size will be determined by the number of patients with intracranial hemorrhage associated with anticoagulation in the clinical records. All electronic medical records that meet the inclusion criteria will be included in the analysis.

Descriptive analysis:

Descriptive statistics will be used for demographic and clinical characteristics of the study sample. This will include measures of central tendency (mean, median) and measures of dispersion (standard deviation, range).

Analytic (Inferential) analysis:

A univariate analysis will take place in order to examine the relationship between demographic and clinical variables with anticoagulation-associated intracranial hemorrhage This will include chi-squared tests for categorical data and T-tests or Mann-Whitney U Tests for continuous data.

A multivariable logistic regression analysis will be done to identify independent predictors of intracranial bleeding associated with anticoagulant therapy. The variables to include in the model will be determined by de univariate analysis results.

The investigators will consider a p-value under 0.05 for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Intracranial hemorrhage diagnosis and concomitant oral anticoagulant therapy
* Available clinical record from January 2015 to July 2023

Exclusion Criteria:

* Non available clinical record
* Patients that did not complete follow up on days 30 and 90 after an intracranial bleeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All outpatients and/or hospitalized patients and patients from the emergency room of the National Institute of Neurology and Neurosurgery Manuel Velasco Suárez with intracranial hemorrhage diagnosis under anticoagulant therapy such as Vitamin K antangonists, Factor Xa inhibitors or direct thrombin inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Know incidence and prevalence of intracranial bleeding events | From January 2015 to November 2023
  To identify the incidence and prevalence of intracranial bleeding events associated to oral anticoagulant therapy including vitamin k antagonists, factor Xa inhibitors and factor 2a inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Vanessa Cano Nigenda, MD, Study Director — Instituto Nacional de Neurología y Neurocirugía. Manuel Velasco Suárez
Locations (1):
- Instituto Nacional de Neurología y Neurocirugía, Mexico City, Mexico

REFERENCES:
- [Result] Adachi T, Hoshino H, Takagi M, Fujioka S; Saiseikai Stroke Research Group. Volume and Characteristics of Intracerebral Hemorrhage with Direct Oral Anticoagulants in Comparison with Warfarin . Cerebrovasc Dis Extra. 2017;7(1):62-71. doi: 10.1159/000462985. Epub 2017 Apr 3. PMID 28376486
- [Result] Ballestri S, Romagnoli E, Arioli D, Coluccio V, Marrazzo A, Athanasiou A, Di Girolamo M, Cappi C, Marietta M, Capitelli M. Risk and Management of Bleeding Complications with Direct Oral Anticoagulants in Patients with Atrial Fibrillation and Venous Thromboembolism: a Narrative Review. Adv Ther. 2023 Jan;40(1):41-66. doi: 10.1007/s12325-022-02333-9. Epub 2022 Oct 16. PMID 36244055
- [Result] Barrios V, Cinza-Sanjurjo S, Gavin O, Egocheaga I, Burgos-Pol R, Soto J, Polanco C, Suarez J, Casado MA. Cost and burden of poor anticoagulation control with vitamin K antagonists in patients with nonvalvular atrial fibrillation in Spain. Rev Esp Cardiol (Engl Ed). 2021 Sep;74(9):773-780. doi: 10.1016/j.rec.2020.06.033. Epub 2020 Sep 24. English, Spanish. PMID 32980294
- [Result] Flaherty ML. Anticoagulant-associated intracerebral hemorrhage. Semin Neurol. 2010 Nov;30(5):565-72. doi: 10.1055/s-0030-1268866. Epub 2011 Jan 4. PMID 21207349
- [Result] Grysiewicz R, Gorelick PB. Incidence, mortality, and risk factors for oral anticoagulant-associated intracranial hemorrhage in patients with atrial fibrillation. J Stroke Cerebrovasc Dis. 2014 Nov-Dec;23(10):2479-2488. doi: 10.1016/j.jstrokecerebrovasdis.2014.06.031. Epub 2014 Oct 29. PMID 25440361
- [Result] Rozjabek HM, Coleman CI, Ashton V, Laliberte F, Oyefesobi P, Lejeune D, Germain G, Schein JR, Yuan Z, Lefebvre P, Peterson ED. Healthcare costs of stroke and major bleeding in patients with atrial fibrillation treated with non-vitamin K antagonist oral anticoagulants. J Med Econ. 2019 Aug;22(8):751-759. doi: 10.1080/13696998.2019.1603156. Epub 2019 Apr 25. PMID 30939954
- [Result] Hellenbart EL, Faulkenberg KD, Finks SW. Evaluation of bleeding in patients receiving direct oral anticoagulants. Vasc Health Risk Manag. 2017 Aug 23;13:325-342. doi: 10.2147/VHRM.S121661. eCollection 2017. PMID 28860793
- [Result] Izumi C, Miyake M, Amano M, Kitai T, Obayashi Y, Takegami M, Kimura T, Sugio K, Matsumoto T, Nishimura K, Furukawa Y. Registry of antithrombotic therapy in atrial fibrillation patients with bioprosthetic valves: A retrospective observational study. J Cardiol. 2020 Jul;76(1):44-50. doi: 10.1016/j.jjcc.2020.02.006. Epub 2020 Mar 7. PMID 32156512
- [Result] Lip GYH, Banerjee A, Boriani G, Chiang CE, Fargo R, Freedman B, Lane DA, Ruff CT, Turakhia M, Werring D, Patel S, Moores L. Antithrombotic Therapy for Atrial Fibrillation: CHEST Guideline and Expert Panel Report. Chest. 2018 Nov;154(5):1121-1201. doi: 10.1016/j.chest.2018.07.040. Epub 2018 Aug 22. PMID 30144419
- [Result] Milling TJ Jr, Frontera J. Exploring indications for the Use of direct oral anticoagulants and the associated risks of major bleeding. Am J Manag Care. 2017 Apr;23(4 Suppl):S67-S80. PMID 28581331
- [Result] Miyamoto S, Ikeda T, Ogawa S, Kitazono T, Nakagawara J, Minematsu K, Murakawa Y, Iwashiro S, Takeichi M, Kidani Y, Okayama Y, Sunaya T, Sato S, Yamanaka S. Clinical Risk Factors of Thromboembolic and Major Bleeding Events for Patients with Atrial Fibrillation Treated with Rivaroxaban in Japan. J Stroke Cerebrovasc Dis. 2020 Apr;29(4):104584. doi: 10.1016/j.jstrokecerebrovasdis.2019.104584. Epub 2020 Jan 23. PMID 31983518
- [Result] Qureshi AI, Mendelow AD, Hanley DF. Intracerebral haemorrhage. Lancet. 2009 May 9;373(9675):1632-44. doi: 10.1016/S0140-6736(09)60371-8. PMID 19427958
- [Result] Rohla M, Weiss TW, Pecen L, Patti G, Siller-Matula JM, Schnabel RB, Schilling R, Kotecha D, Lucerna M, Huber K, De Caterina R, Kirchhof P. Risk factors for thromboembolic and bleeding events in anticoagulated patients with atrial fibrillation: the prospective, multicentre observational PREvention oF thromboembolic events - European Registry in Atrial Fibrillation (PREFER in AF). BMJ Open. 2019 Mar 30;9(3):e022478. doi: 10.1136/bmjopen-2018-022478. PMID 30928922
- [Result] Roskell NS, Samuel M, Noack H, Monz BU. Major bleeding in patients with atrial fibrillation receiving vitamin K antagonists: a systematic review of randomized and observational studies. Europace. 2013 Jun;15(6):787-97. doi: 10.1093/europace/eut001. Epub 2013 Feb 13. PMID 23407628
- [Result] Ruiz-Sandoval JL, Chiquete E, Garate-Carrillo A, Ochoa-Guzman A, Arauz A, Leon-Jimenez C, Carrillo-Loza K, Murillo-Bonilla LM, Villarreal-Careaga J, Barinagarrementeria F, Cantu-Brito C; RENAMEVASC investigators. Spontaneous intracerebral hemorrhage in Mexico: results from a Multicenter Nationwide Hospital-based Registry on Cerebrovascular Disease (RENAMEVASC). Rev Neurol. 2011 Dec 16;53(12):705-12. English, Spanish. PMID 22127656
- [Result] Deitelzweig S, Neuman WR, Lingohr-Smith M, Menges B, Lin J. Incremental economic burden associated with major bleeding among atrial fibrillation patients treated with factor Xa inhibitors. J Med Econ. 2017 Dec;20(12):1217-1223. doi: 10.1080/13696998.2017.1362412. Epub 2017 Aug 11. PMID 28760063
- [Result] You JJ, Singer DE, Howard PA, Lane DA, Eckman MH, Fang MC, Hylek EM, Schulman S, Go AS, Hughes M, Spencer FA, Manning WJ, Halperin JL, Lip GYH. Antithrombotic therapy for atrial fibrillation: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e531S-e575S. doi: 10.1378/chest.11-2304. PMID 22315271